CLINICAL TRIAL: NCT04816045
Title: Neoadjuvant Electrochemotherapy for Colorectal Cancer - a Randomized Controlled Trial
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-032-2020
Record Dates: First submitted 2021-02-24; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Electroporation; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients and investigators are blinded. The allocation list is located at the pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Electrochemotherapy with bleomycin
  Interventions: Procedure: Electrochemotheraoy
- Control (Active Comparator): Electroporation with saline
  Interventions: Procedure: Electroporation with saline (placebo)

INTERVENTIONS:
Procedure: Electrochemotheraoy — Electrochemotherapy (ECT) is endoscopic electroporation in combination with bleomycin
  Arms: Intervention
Procedure: Electroporation with saline (placebo) — Electroporation in the control group is performed endoscopically with saline
  Arms: Control

SUMMARY:
This is a randomized controlled trial investigating efficacy of electrochemotherapy for early colorectal cancer

DETAILED DESCRIPTION:
This is a phase 2 randomized controlled trial. The study is blinded. The aim of this study is to establish the safety and efficacy of treating patients with early colorectal cancer with electrochemotherapy, compared with electroporation alone, as a down staging and immune-response enhancing treatment prior to intended curative surgery. The study involves recruitment of patients with histologically verified rectal and sigmoid colon cancer with no indication for neoadjuvant chemoradiotherapy (experimental or standard care based) prior to intended curative surgery. In total the study will involve 24 patients, of these, 12 patients are treated with electrochemotherapy (bleomycin) and 12 patients with electroporation alone (placebo)

In relation to the intervention, clinical examination, blood samples, biopsies and questionnaires will be collected to evaluate safety, tumor respons and immunologic response to the treatment.

Patients will be followed for one month after the elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be mentally capable of understanding the information given.
* Patients must give written informed consent.
* Endoscopically suspected or histologically verified malignant tumor of the rectum or sigmoid colon.
* Tumor described as passable at index endoscopy.
* Men or women aged at least 18 years.
* Case reviewed by MDT (surgery, radiology, oncology). Case considered curable with standard surgical resection.
* ASA class I-II (Classification of the American Society of Anesthesiology)

Exclusion Criteria:

* Indication for neoadjuvant chemoradiation or chemotherapy prior to surgery
* Uncorrectable coagulation disorder.
* Patients with ICD or pacemaker units.
* Ongoing immunosuppressive treatment.
* Patients with concomitant use of phenytoin.
* Myocardial insufficiency, defined as NYHA class >2
* Concurrent treatment with an investigational medicinal product.
* Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study recruitments.
* Advanced tumor stages, clinical UICC stage IV.
* Acute surgical resection.
* Pregnancy
* Medical history of severe pulmonary disease.
* Previous cumulative dose of bleomycin exceeding 250mg/m2.
* BMI > 35
* Renal impairment, defined as eGFR <40 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Tumor stage | 6 months
  Preoperative tumor stage will be compared with pathological assessment of the surgical specimen and comared between the two study arms using TNM stage

SECONDARY OUTCOMES:
Gene expressional changes in the tumor microenvironment | 6 months
  Biopises are collected before the intervention and compared with the surgical specimen using NanoString technology. The PanCancer IO 360 gene panel will be used, a predefined panel of 770 genes.
Composition of fusobacterium | 6 months
  To characterize the spatial distribution and organization of bacteria in situ, some of the samples will be assessed microscopically. Confocal laser scanning microscopy will be performed on formalin-fixed, paraffin-embedded tissue of both diseased and normal tissue. This will allow us to investigate treatment affects the bacterial composition of fusobacterium.
PD-1/PD-L1 | 6 months
  Immunohistochemical staining for PD-1/PD-L1
CD3 | 6 months
  Immunohistochemical staining for CD3
CD8 | 6 months
  Immunohistochemical staining for CD8
CD28 | 6 months
  Immunohistochemical staining for CD28
VAR2 | 6 months
  Immunohistochemical staining for VAR2

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, DMSc, Principal Investigator — Zealand University Hospital